CLINICAL TRIAL: NCT00870428
Title: The Predictive Use of Spot Urine Protein/Creatinine Ratios and Decreased Sample Collection Time in the Diagnosis of Preeclampsia
Brief Title: Predicitve Use of Spot Urine Protein/Creatinine Ratios in Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MemorialCare (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Deborah A. Wing, Univeristy of California Irvine
Other Study IDs: 584-08
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; proteinuria
MeSH Terms: conditions — Pre-Eclampsia; Proteinuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preeclampsia Evaluation: Patients who are admitted for the evaluation of preeclampsia

SUMMARY:
The investigators intend to perform a large prospective study looking at the predictability of the random urine protein-to-creatinine ratio compared to the gold standard 24-hour urine protein collection. Furthermore, the investigators plan to investigate whether analysis of proteinuria at shorter time intervals (4 and 8 hours) within the overall 24-hour collection period is predictive of the 24-hour sample. Lastly, the investigators plan to determine whether a combination of the random test with a shorter collection interval is comparable to the 24-hour collection.

DETAILED DESCRIPTION:
Preeclampsia affects approximately 5-8% of pregnancies in the United States with approximately 10% occurring before 34 weeks gestation. The diagnosis of preeclampsia is determined by the presence of hypertension with proteinuria after 20 weeks gestation. The gold standard for measuring proteinuria is a 24-h urine collection for total protein. In the non-pregnant patient, a random urinary protein-to-creatinine ratio has been shown to be a reliable indicator of significant proteinuria. The reliability of this test remains unclear in the pregnant population. Because there are relatively few studies in the pregnant population and many of these studies were poorly designed, limited by sample size, or confounded by other variables, further research in this area is still necessary. The purpose of this study is to determine if there are alternative diagnostic tools for the quantification of total protein excretion in 24-hours to aid in the diagnosis of preeclampsia that can be performed more quickly and efficiently than the gold standard 24-hour urine collection. We intend to perform a large prospective study looking at the predictability of the random urine protein-to-creatinine ratio compared to the gold standard 24-h urine protein collection. Furthermore, we plan to investigate whether analysis of proteinuria at shorter time intervals (4 and 8 hours) within the overall 24-h collection period is predictive of the 24-h sample. Lastly, we plan to determine whether a combination of the random test with a shorter collection interval is comparable to the 24-h collection. The goal would be to make the diagnosis of preeclampsia in a more timely fashion to aid in the prevention of maternal and neonatal morbidity and mortality including eclampsia, HELLP syndrome, acute renal failure, pulmonary edema, DIC, IUGR, IUFD, intracranial bleeding and stroke, Additionally, an earlier diagnosis could also impact patient care by reducing hospital stay, nursing demands, and eliminating the need for cumbersome and likely inaccurate patient 24-h home collections.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over the age of 18 between 24-42 weeks who are being evaluated for preeclampsia with a 24 hour urine protein

Exclusion Criteria:

* Patients with pre-existing proteinuria (>300mg)
* Renal disease
* Evidence of a current or recent (within two weeks of admission) urinary tract infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women between 24-42 weeks who are being evaluated for preeclampsia.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2009-03

PRIMARY OUTCOMES:
To determine if protein excretion determined by spot urine protein-to-creatinine ratios are equivalent to the gold standard 24-h urine protein collections. | 24 hours

SECONDARY OUTCOMES:
To see if total protein excretion obtained from shorter timed urine collections of 4- and 8-hours duration or a combination of the two tests are equivalent to a 24-h urine collection. | 4 hr, 8 hr, 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Wing, MD, Principal Investigator — Univeristy of California Irvine
Locations (1):
- Long Beach Memorial Womens Pavillion, Long Beach, California, United States